CLINICAL TRIAL: NCT05922072
Title: Comparison of Different Preoperative Fasting Times in Pediatric Patients Undergoing Elective General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fatima Numeri, Assistant Professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KingEdwarMU
Record Dates: First submitted 2023-03-07; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Aspiration of Gastric Contents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Intervention Model Description: Total 120 patients will be randomly allocated into two groups using computerized generated numbers (60 in each group). Group A with 6,4 and 2 hours NPO for solids/ formula milk, breast milk and clear fluid respectively. Group B with 6,4 and 1-hour NPO for solids/ formula milk, breast milk and clear fluid respectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long NPO group (Active Comparator): 6,4 and 2 hours NPO for solids/ formula milk, breast milk and clear fluid respectively
  Interventions: Procedure: Nasogastric aspiration for measurement of Residual Gastric Volume; Procedure: Nasogastric Aspiration for Measurement of Gastric pH
- Short NPO group (Experimental): 6,4 and 1-hour NPO for solids/ formula milk, breast milk and clear fluid respectively
  Interventions: Procedure: Nasogastric aspiration for measurement of Residual Gastric Volume; Procedure: Nasogastric Aspiration for Measurement of Gastric pH

INTERVENTIONS:
Procedure: Nasogastric aspiration for measurement of Residual Gastric Volume — The patients enrolled in this study undergoing elective general anesthesia,their mean gastric residual volume will be measured by taking Nasogastric tube aspirate.
Procedure: Nasogastric Aspiration for Measurement of Gastric pH — The patients enrolled in this study undergoing elective general anesthesia,their mean gastric gastric PH will be measured by taking Nasogastric tube aspirate.

SUMMARY:
Rationale of this study is to provide an evidence on minimal safe clear fluid fasting duration without the risk of aspiration of gastric contents during elective pediatric procedures under general anesthesia.

DETAILED DESCRIPTION:
Pre-operative fasting is a specific time period before a procedure in which participants will be advised not to take any liquid or solid by mouth. Nil per oral (NPO) is a universally accepted practice before elective general anesthesia in order to reduce gastric contents aspiration. In the period of chloroform anesthesia NPO was introduced because of vomiting and discomfort associated with anesthesia. Hence prevention from aspiration of gastric contents was a main focus during general anesthesia. With introduction of better anesthesia drugs recommendations were given to keep minimal fasting time before general anesthesia.

Recent guidelines suggest six, four and two hours fasting for solids/ infant formula milk, breast milk and clear fluids respectively. It is common practice to keep children NPO for 6 hours before surgery. But many times, children have to suffer excessive unnecessary fasting due to delayed surgery that lead to reduction in systolic blood pressure, induce catabolic state and behavioral effects. Moreover prolonged fasting increases insulin resistance and may increase the inflammatory response to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients
2. Age between 1 to 12 years
3. Patients undergoing elective surgical procedures ( orchidopexy, lymph node biopsy, skin grafting, tongue ties and hernia repair ) under general anesthesia

Exclusion Criteria:

1.Patients with co-morbidities like acid peptic disease with history of dyspepsia and family history or self-history of diabetes mellitus.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Mean residual gastric volume | 6 Months
  Mean Residual Gastric Volume will be measured in mililiter

SECONDARY OUTCOMES:
Gastric pH | 6 months
  Gastric pH will be measured by pH Litmus paper

CONTACTS AND LOCATIONS:
Locations (1):
- Paeds Surgery Department Mayo Hospital, Lahore, Punjab Province, Pakistan